CLINICAL TRIAL: NCT03727178
Title: Acute Acromioclavicular Dislocation: Epidemiology, Natural History and Analysis of Prognostic Factors
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristine Bramsen Andersen, Medical Doctor, Hvidovre University Hospital
Other Study IDs: AC_lux_cohort
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: Acromioclavicular Joint Dislocation; AC joint dislocation; Treatment; Conservative treatment; Type III AC dislocation; Grade III AC dislocation; AC joint; Rockwood; Rockwood type III; Rockwood grade III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim:

To evaluate non-operative treatment of acute acromioclavicular (AC) joint dislocation and define prognostic factors to guide the choice of treatment in order to develop an individualized treatment algorithm.

Objectives:

1. To investigate whether a sub classification of Rockwoods type III in a stable type IIIA and an unstable type IIIB, as suggested by ISAKOS (International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine), is clinically relevant. Clinically relevant is defined as a difference in the WOSI score of >14%
2. To evaluate clinical, functional and radiological results, along with patient-reported health, 6 weeks, 3 months, 6 months and 1 year after acute AC dislocation
3. To investigate whether specific factors are of prognostic value to the result after non-operative management of acute AC dislocation
4. To investigate if Rockwoods classification of AC dislocations is of prognostic value for the rehabilitation after the injury.

Type of study: Prospective cohort study. 100 patients will be included.

Time schedule:

Recruitment of patients is planned to begin November 2018. It is expected that the inclusion will span 1 year, provided an average of 2 patients included per week. With a 1-year follow-up for each patient the total study period is expected to be 2 years.

Set-up:

In the Capital Region of Denmark the majority of patients with acute AC joint dislocation are treated non-operatively. A collar'n cuff is applied in the emergency room and the patient is instructed to begin non-weight bearing exercises after 1-3 weeks.

100 patients with acute AC-joint dislocation will be included in the cohort and evaluated at controls 6 weeks, 3 months, 6 months and 1 year after the injury. The patients will be identified from X-rays obtained in the Emergency Departments at three Danish Hospitals.

At each control the patient will reply to 2 questionnaires regarding their shoulder-related function and quality of life, be evaluated through 5 clinical tests, and 2 different X-rays of the AC-joint will be obtained.

DETAILED DESCRIPTION:
Introduction:

Acromioclavicular (AC) joint dislocations are common injuries accounting for 9-12% of all injuries to the shoulder girdle. The injuries are graded according to Rockwoods classification type I-VI. There is consensus on the treatment of Rockwood type I and II which rehabilitates well with conservative treatment, and for high-grade injuries of types IV, V and VI, which usually requires surgery. However the treatment of the most common type, type III, has remained controversial for the last 30 years. To assess this problem, ISAKOS (International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine) Upper Extremity Committee in 2014 provided a modified Rockwood classification, suggesting a sub-classification of the debated type III in a stable type IIIA and an unstable type IIIB.

The purpose of this sub-classification is to identify and differentiate patients, who are expected to rehabilitate well with conservative treatment from those who would benefit from early surgical intervention, i.e. type IIIA and IIIB. Type IIIA is considered stable and is characterized by absence of scapula dyskinesia and no overriding of the clavicle to acromion. Type IIIB is characterized by presence of scapula dyskinesia and no overriding of the clavicle to acromion.

Aim:

To evaluate non-operative treatment of acute acromioclavicular (AC) joint dislocation and define prognostic factors to guide the choice of treatment in order to develop an individualized treatment algorithm.

Objectives:

1. To investigate whether a sub classification of Rockwoods type III in a stable type IIIA and an unstable type IIIB, as suggested by ISAKOS, is clinically relevant. Clinically relevant is defined as a difference in the WOSI score of >14%
2. To evaluate clinical, functional and radiological results, along with patient-reported health, 6 weeks, 3 months, 6 months and 1 year after acute AC dislocation
3. To investigate whether specific factors are of prognostic value to the result after non-operative management of acute AC dislocation
4. To investigate if Rockwoods classification of AC dislocations is of prognostic value for the rehabilitation after the injury.

Study design: The study is carried out as a prospective cohort study. 100 patients will be included.

Time schedule:

Recruitment of patients for the study is planned to begin in November 2018. It is expected that the inclusion will span 1 year, provided an average of 2 patients included per week. With a 1-year follow-up for each patient the total study period is expected to be 2 years.

Methods:

Recruitment:

100 patients with acute AC-joint dislocation from the Emergency Departments at three different hospitals in the Capital Region of Denmark (Hvidovre, Glostrup and Amager hospitals) will be included in the cohort. Patients with superior displacement of the clavicle to the acromion are of interest to the study.

At the Emergency Departments, the patients will receive the standard conservative treatment of collar'n cuff for 1-3 weeks.

To identify patients, all X-rays of the AC-joint and the clavicle obtained at the three hospitals will be evaluated weekly, identifying the presence and degree of potential AC dislocations. If the patient meet the inclusion criterias, he or she will be invited to participate in the cohort.

Follow-up:

Participants will be offered an appointment in the ambulatory for baseline evaluation. Follow-up measurements will be performed at 6 weeks, 3 months, 6 months and 1 year after the injury. The study's primary endpoint is at the 3 month mark.

At the follow-ups, participants will be evaluated clinically, functionally and radiologically. Primary outcome measure is the patient's self-reported shoulder-related quality of life, evaluated using WOSI (Western Ontario Shoulder Instability Index). As secondary outcomes patients will evaluate their functional limitations and pain with SPADI (Shoulder Pain and Disability Index), the cosmetic results with NRS (Numeric Rating Scale) and attend a clinical evaluation regarding range of motion (ROM), the presence of scapular dyskinesia, antero-posterior/superior-inferior instability of the clavicle and O'Briens test. Two radiographs of the AC-joint will be obtained to determine the coraco-clavicular distance as well as the degree of overriding of the clavicle to acromion.

It is expected that a number of patients in the cohort, due to sustainable pain and non-acceptable disability, will be offered surgical treatment. This group will be followed exactly like the group of conservatively treated patients. The two groups will be compared both according to their demographical data and their outcome.

Discontinuation:

Each patient can choose to withdraw from the trial at any time. A patient may also be withdrawn from the trial at any time based on the investigators' discretion.

Data Registration:

All relevant data is recorded and stored in a specially designed database; RedCap. The data registration has been approved by the Danish Data Protection Agency and The Ethical committee of the Capital Region of Denmark.

Statistics:

The cohort will be described descriptively regarding demographic parameters as well as primary and secondary outcomes. The change of the outcomes over time will be described using relevant statistics according to the characteristics of the variables and if necessary the normal distribution. A regression analysis will be used to evaluate the association between prognostic factors and recovery.

Sample size:

The sample size is calculated to detect if a clinical relevant difference in WOSI-score exists between a group with stable (type IIIA) and unstable (type IIIB) AC dislocations. The calculation is based on a clinical relevant difference in WOSI-score of 14%, a standard deviation, SD, of 20%, a significance level of 0,05 and a power of 90%. According to this calculation the study demands 88 patients but because of the risk of drop-out, 100 patients will be included.

Ethical considerations:

The project is approved by the National Committee on Health Research Ethics. The purpose of the study is to follow the natural history of a common injury, where guidelines for the treatment already exist. There is no intervention in the study - patients enrolled will receive the standard treatment in the Emergency Departments. They will be offered standardized physiotherapy and extra controls, which is considered an advantage for the patients as they receive a thorough follow-up and examination of the healing process. The disadvantages for the patients are: 1) Participation in the study is time-consuming: Patients need to attend 4 extra controls, each lasting approximately 1h. 2) Exposure to radiation: At each control, 2 x-rays of the shoulder will be obtained. However the radiation exposure is very small, only 0,1-0,3 mSv/ x-ray, equivalent to a few weeks of background radiation. It is believed that the potential benefits for both patients in the study and future patients with AC dislocations (thorough follow-up and individualized treatment,) exceed the the potential inconveniences (additional follow-up audits and light exposure to radiation).

ELIGIBILITY:
Inclusion Criteria:

1. Trauma to the shoulder and pain from the AC joint within the last 7 days.
2. X-ray from the Emergency Room revealing >50% superior displacement of the lateral tip of the clavicle to acromion.
3. Age 18-60 years
4. The patient must be expected to be able to attend rehabilitation and post- examinations.
5. The patient must be able to speak and understand Danish
6. Signed informed consent.

Exclusion Criteria:

1. History of previous AC joint dislocation or shoulder trauma (ipsi/contralateral)
2. Fracture to the upper extremity at time of injury.
3. Associated injuries to the upper extremity causing limitation of function, including fracture or dislocation of the shoulder

3) Terminal illness or severe medical illness. ASA (American Society of Anesthesiologists) group ≥ 3

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients with acute acromioclavicular dislocation, admitted to the Emergency departments at Hvidovre, Glostrup and Amager Hospitals (Copenhagen). All patients will be treated according the standard regimen.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability score (WOSI) in percentage | 3 months
  The WOSI score is a Patient Reported Outcome Measure (PROM) evaluating disease-specific quality of life patients with shoulder instability, but can also be used for evaluation of other injuries to the shoulder girdle. In the questionnaire the patients answer 21 questions according to 4 different domains: physical function, sports/recreation/work, lifestyle and emotional well-being. Each question is scored 1-100 points by marking on a visual analog scale (VAS), and the summation of all the questions results in a final WOSI score, ranging from 0-2100, where 0 is the best score with no influence on quality of life and 2100 is the worst score with the patient experiencing extreme distress in shoulder-related quality of life. The score is often transferred into a %-score, where 100% is best and 0% is worst. The minimal clinically important difference is reported to be 14%. The score will be used as a measurement to determine how well the patients are doing throughout the follow-up period.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline, 6 weeks, 3 months, 6 months, 1 year
  SPADI is a measurement (a PROM) designed to evaluate patient-reported pain and shoulder disability. For each question, the patient marks his answer on a 0-10 numerical rating scale, where 0 is "no pain" or "no disability" and 10 is "worst pain" or "maximal disability". The total score is expressed as percentage, 0-100%, where a lower score equals a better result. The minimal clinically important difference is 8%.
Western Ontario Shoulder Instability score (WOSI) in percentage | Baseline, 6 weeks, 6 months, 1 year
  The WOSI score is a Patient Reported Outcome Measure (PROM) evaluating disease-specific quality of life patients with shoulder instability, but can also be used for evaluation of other injuries to the shoulder girdle. In the questionnaire the patients answer 21 questions according to 4 different domains: physical function, sports/recreation/work, lifestyle and emotional well-being. Each question is scored 1-100 points by marking on a visual analog scale (VAS), and the summation of all the questions results in a final WOSI score, ranging from 0-2100, where 0 is the best score with no influence on quality of life and 2100 is the worst score with the patient experiencing extreme distress in shoulder-related quality of life. The score is often transferred into a %-score, where 100% is best and 0% is worst. The minimal clinically important difference is reported to be 14%. The score will be used as a measurement to determine how well the patients are doing throughout the follow-up period.
The patient's satisfaction with the cosmetic result | Baseline, 6 weeks, 3 months, 6 months, 1 year
  On a scale from 0 to 10, where 0 is very dissatisfied and 10 is very satisfied
Return to work: Number of days passed from the day of the injury to the day where the patient resume his work. | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Number of days passed from the day of the injury to the day where the patient resume his work.
Return to sports: Number of days passed from the day of the injury to the day where the patient resume his sports. | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Number of days passed from the day of the injury to the day where the patient resume his sports.
Range of motion: Bilateral active flexion, measured in degrees. | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Bilateral active flexion of the shoulders, measured in degrees.
Range of motion: Bilateral active abduction, measured in degrees. | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Bilateral active abduction of the shoulders, measured in degrees.

OTHER OUTCOMES:
Scapula dyskinesis | 6 weeks, 3 months, 6 months, 1 year
  Scapula dyskinesia is defined as abnormal movement, asymmetry or "winging" of the shoulder blade with the patient performing 5x bilateral shoulder flexion followed by 5x bilateral shoulder abduction. If scapula dyskinesia is present in any of the movements, the test is considered positive.
Antero-posterior instability | 6 weeks, 3 months, 6 months, 1 year
  With one hand, the examiner fixates the acromion, while the stability of the joint is tested in the horizontal plane by moving the distal tip of the clavicle antero-posteriorly. The test is positive if there is more movement on the affected side
Superior-inferior instability | 6 weeks, 3 months, 6 months, 1 year
  The stability of the joint in the vertical plane is tested by pressing the protruding lateral tip of the clavicle up and down. The non-affected side is used as a control
O'Briens test | 6 weeks, 3 months, 6 months, 1 year
  With the patient standing or sitting, the shoulder is placed in a 90° flexed and 10-15° horizontally adducted position. In this position, and with the arm stretched, the patient fully internally rotates the shoulder causing the little finger to point upwards. The examiner then applies a distal stabilizing force as the patient is instructed to apply an upward force, causing stress to the AC-joint. The patient will then be asked to perform the same procedure, but with the thump pointing upwards. The test is considered positive if any part of the test results in pain or clicking in the shoulder.
The coraco-clavicular distance expressed in percentage compared to the non-affected side | Baseline, 6 weeks, 3 months, 6 months, 1 year
  Bilateral Zanca provides the best possible visualization of the AC-joint. The coraco-clavicular distance will be measured and expressed in percentage compared to the non-affected side.
Positive Basamani: overriding of the distal tip of the clavicle to acromion | Baseline, 6 weeks, 3 months, 6 months, 1 year
  The Basamani (cross body adduction) view is obtained with the patients' arm in a cross-over position. This will stress the acromioclavicular joint and reveal a potential overriding of the clavicle to acromion - which might be significant for an unstable joint.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine B Andersen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Copenhagen, Denmark